CLINICAL TRIAL: NCT00142571
Title: Ph III Random Trial of 120-Min Infusion Gemcitabine v. 90-Min Infusion Gemcitabine + Docetaxel in Unresectable Soft Tissue Sarcoma: A Multi-Disciplinary Trial of the North Amer. Sarcoma Study Group of the Connective Tissue Oncology Society
Brief Title: Comparison of Gemcitabine v. Gemcitabine Plus Docetaxel in Unresectable Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Connective Tissue Oncology Society (Other); M.D. Anderson Cancer Center (Other); Massachusetts General Hospital (Other); Mayo Clinic (Other); University of Michigan Rogel Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-129
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-10

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; Gemcitabine; Docetaxel
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel

INTERVENTIONS:
Drug: Gemcitabine
Drug: Docetaxel

SUMMARY:
The purpose of this study is to compare the drug gemcitabine to two drugs, gemcitabine and docetaxel, to find out which treatment is better for people with sarcomas.

DETAILED DESCRIPTION:
This research is being done because better treatments for sarcomas are needed. This is a phase III study. This means that one treatment is being compared to another to find out which is better. We are comparing the drug gemcitabine to the two drugs gemcitabine and docetaxel to find out which treatment is better for people who have sarcomas. From previous studies we know that gemcitabine causes shrinking of some people's sarcoma tumors. We also know that gemcitabine and docetaxel are useful for sarcomas as well, but we believe the two drugs together may be more toxic than the single drug alone. In this study we are trying to answer the question: "Is the combination of gemcitabine and docetaxel any better than just gemcitabine alone?"

This is a randomized Phase III trial comparing two treatment regimens in patients with unresectable soft tissue sarcoma. The failure rates observed on both treatment arms (failure defined as progression or death) will be compared to determine which regimen results in the lowest failure rate (Primary objective). As a secondary endpoint, the percentage of patients who are failure-free (failure defined as progression or death) at 3 months and 6 months will be compared between the two arms (Secondary objective).

This trial, sponsored by the North American Sarcoma Study Group of the Connective Tissue Oncology Society, is being done at a number of hospitals around the country and is expected to enroll up to 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven soft tissue sarcoma (except the following histologies: gastrointestinal stromal tumors (GIST), Kaposi's Sarcoma, mesotheliomas
* Age >= 10 years
* Recurrent or progressive disease defined as an increase in size of any existing tumor mass, or the development of new tumor mass or masses, which is not amenable to definitive surgical therapy.
* Patients may have had another cancer but there must be convincing clinical evidence that the sarcoma is the disease requiring therapeutic intervention. (ie. Several sarcoma patients have had had a prior cancer (Hodgkin's disease or breast cancer) treated years previously and then developed a clinically active sarcoma.)
* Patients may have failed no more than 3 prior chemotherapy regimens.
* Measurable disease as defined by RECIST. Measurable disease is the presence of at least one measurable lesion. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. A measurable lesion is one that can be accurately measured in at least one dimension with longest diameter >20 mm using conventional techniques or >10 mm with spiral CT scan.
* Karnofsky performance status of greater than or equal to 60%
* Peripheral neuropathy, if present, must be < or = to grade 1
* At least 3 weeks since prior chemotherapy (10 days if the patient was on imatinib, thalidomide, or an interferon)
* At least 3 weeks since prior radiation therapy
* Absolute neutrophil count > 1,500/mm3
* Hemoglobin > 8.0 g/dl
* Platelet count > 100,000/mm3
* Total Bilirubin < upper limit of normal (ULN).
* ALT (SGOT) or AST (SGPT) <5 x ULN.
* Alkaline Phosphatase < 2.5 x ULN.
* Serum creatinine < or equal to 2.0 mg/dL
* Women of child-bearing potential must have a negative serum pregnancy test
* Men and women of child-bearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter (approximately 3 months)
* If the patient is 18 or older, the patient must be capable of providing written, informed consent. If the patient is younger than 18, written and voluntary informed consent from patient's parents or legal guardians and the patient's assent are required.

Exclusion Criteria:

* Soft tissue sarcomas with the following histologies: gastrointestinal stromal tumors (GIST), Kaposi's sarcoma, mesotheliomas
* Active or uncontrolled infection (on antibiotic therapy for acute or chronic infection)
* Prior treatment with gemcitabine or docetaxel
* Peripheral neuropathy > or = grade 2
* History of known hypersensitivity reaction to agents formulated in polysorbate 80, the solubilizing agent for docetaxel [e.g. interferon alpha-2a, children's ibuprofen suspension (Advil), terconazole (Terazol), lamivudine (Epivir), etoposide, amiodarone, vaccines (DtaP, influenza), bupropion (Wellbutrin), Vitamins B12, C+zinc+selenium].
* Uncontrolled, central nervous system metastases

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2003-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine whether the failure rate (defined as progression or death) among patients with unresectable soft tissue sarcoma is improved with gemcitabine plus docetaxel compared with gemcitabine alone

SECONDARY OUTCOMES:
Determine whether the failure rate (defined as progression or death) at 3 and 6 months is improved among patients with unresectable soft tissue sarcoma treated with gemcitabine plus docetaxel compared with those treated with gemcitabine alone.
Overall survival will be evaluated
Response rate will be evaluated
Toxicity will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://mskcc.org